CLINICAL TRIAL: NCT05813171
Title: The Effects of Dietary Supplementation Allicor on Patients With Multifocal Atherosclerosis After Peripheral Artery Revascularization Treatment During a Year
Brief Title: The Effects of Allicor on Patients After Revascularization Treatment During a Year
Acronym: TEA-PARTY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute for Atherosclerosis Research, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IAR-AL-MFA
Record Dates: First submitted 2023-04-02; First posted 2023-04-14 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Atherosclerosis; Peripheral Arterial Disease
Keywords: atherosclerosis; inflammation; DNA, Mitochondrial
MeSH Terms: conditions — Atherosclerosis; Peripheral Arterial Disease; Inflammation | interventions — tebufenozide

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with two parallel groups of participants
Who Masked: Participant, Care Provider
Masking Description: A randomized, double-blinded, placebo-controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Allicor (Active Comparator): Dietary Supplement: Allicor 150 mg capsule by mouth two times a day during the year
  Interventions: Dietary Supplement: Allicor
- Placebo (Placebo Comparator): Placebo capsule manufactured to mimic Allicor 150 mg capsule by mouth two times a day during the year
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Allicor — Participants will take Allicor capsules in addition to standard treatment for a year.
  Other Names: 150 mg capsules of dried dried garlic powder
  Arms: Experimental: Allicor
Drug: Placebo — Participants will take the placebo capsules in addition to standard treatment for a year.
  Other Names: 150 mg inert capsules mimic capsules Allicor
  Arms: Placebo

SUMMARY:
A significant challenge in medical care is atherosclerotic occlusion of peripheral arteries, such as lower extremities and brachiocephalic arteries, which can eventually lead to loss of limbs or fatal ischemic strokes. Revascularizing surgical interventions can restore the lumen of the arteries and provide an effective way to treat such patients. However, up to a third of patients need re-intervention or experience cardiovascular complications within a year after surgery. The purpose of this study is to evaluate the effect of adding the natural dietary supplement Allicor to conventional treatment on the incidence of cardiovascular complications and treatment effectiveness 12 months after revascularization. Another valuable area of investigation is the search for predictors of long-term cardiovascular complications after revascularization, which could be markers of inflammation and heteroplasmy levels in the patient's mitochondrial genome.

DETAILED DESCRIPTION:
Recently, atherosclerosis of large arteries has become a common problem affecting the quality of life and life expectancy of the population. In addition to atherosclerosis of coronary arteries leading to myocardial ischemia, another significant issue is atherosclerosis of the lower limb and brachiocephalic arteries. Typically, arteries are affected in multiple areas, resulting in multifocal atherosclerosis of several arterial basins. Consequently, 14 to 19% of patients suffering from damage to the arteries of the lower extremities have significant stenosis of the common carotid arteries. Clinical guidelines from the European Society of Cardiology (ESC) and the European Society for Vascular Surgery (ESVS) emphasize the need to examine other arteries in patients with atherosclerosis of the arteries of the lower extremities. Clinical screening for carotid and subclavian artery stenosis is also recommended.

The surgical method for treating arterial occlusive lesions includes revascularization interventions to restore blood flow, thus eliminating tissue ischemia and preventing fatal and disabling consequences. In addition to surgical treatment, medications that lower blood cholesterol and reduce blood thrombogenesis are used.

An important predictor of disease and treatment efficiency is the level of systemic inflammatory markers, such as protein-C. An anti-inflammatory approach is not used for treating patients with multifocal atherosclerosis. However, investigating new markers of inflammation may be promising for the development of new diagnostics.

Insofar as up to a third of patients face the need for re-intervention or suffer cardiovascular complications within a year after revascularization surgery, the search for new approaches to treat multifocal arterial atherosclerosis is necessary.

Long-term use of drugs of natural origin with anti-inflammatory and anti-atherosclerotic effects may be promising.

Dietary Supplementation Allicor consists of dried garlic. There is a trial study (ClinicalTrials.gov Identifier: NCT01734707) that determined the ability of Allicor to have a beneficial effect on patients with atherosclerosis, and there are also data on the beneficial effect of Allicor on the condition of patients with coronary heart disease. Another randomized, double-blind, placebo-controlled trial of a dietary supplement made of garlic (ClinicalTrials.gov Identifier: NCT03860350) found benefits for patients with coronary artery atherosclerosis. Thus, there is reason to believe that Allicor will improve treatment outcomes in patients with multifocal atherosclerosis.

The aim of this study is to investigate how the addition of Allicor to the standard treatment affects the incidence of serious cardiovascular events during a year after revascularization intervention. Also to be assessed is the need for repeated operations, as well as an evaluation of arterial flow and arterial wall. The study will also assess promising markers related to atherosclerosis and inflammation - an in vitro monocyte cytokine release test, and heteroplasmy levels of the patient's mitochondrial genome variants associated with atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age >40 and <75 years
2. A revascularization (including stenting, endarterectomy, artery prosthetic or bypass grafting) is indicated for the patient because of chronic atherosclerotic obliteration of the arteries of the lower extremities and/or common carotid arteries.
3. Patients passed a complex of instrumental and laboratory examinations before revascularization, including X-ray contrast angiography or ultrasound examination of common carotid arteries and arteries of the lower extremities, the ankle-brachial index (ABI) assessment, biochemical analysis of blood included assessment of cholesterol, triglycerides, low density lipoproteins, high density lipoproteins and glucose levels.
4. The possibility of monitoring the patient for 12 months after revascularization, including phone contacts and visits to the clinic after 6 and 12 months.
5. Patient or legal authorized representative capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Repeated revascularization surgery.
2. Trophic ulcers of the lower extremities.
3. Critical and urgent cardiovascular conditions: tissue ischemia stage III-IV, stroke, acute coronary syndrome, myocardial infarction, chronic heart failure III and IV class NYHA (New York Heart Association).
4. Other critical and urgent conditions not associated with cardiovascular diseases, including the need for urgent interventions, chronic renal failure stages IV-V (creatinine clearance < 30 ml / min according to the Cockcroft-Gault Equation)
5. High degree of disability of the patient (4 or higher points on the modified Rankin scale).
6. History of systemic autoimmune diseases.
7. Significant weight loss (> 10% of body weight in the previous year) of unknown etiology.
8. Conditions that limit adherence to participation in the study (dementia, neuropsychiatric diseases, drug addiction, alcoholism, etc.).
9. Participation in other clinical studies (or use of investigational substances) within 3 months prior to study entry.
10. Patients with malignant tumors, including the postoperative period with chemotherapy and/or radiation therapy.
11. Carriers of HIV or viral hepatitis
12. Pregnancy or breast feeding
13. Refusal to participate in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of fatal cardiovascular events | Evaluated in 12 months from revascularization interventions
  Fatal cardiovascular events include: death from myocardial infarction, other forms of coronary heart disease (CHD), stroke, including sudden death and death within 24 hours of symptom onset, death from other non-coronary cardiovascular diseases except definitely non-atherosclerotic causes of death.
Frequency of clinically significant cardiovascular events | Evaluated in 12 months from revascularization interventions
  Clinically significant cardiovascular events include: acute myocardial infarction and acute coronary syndrome, acute cerebrovascular accident, progressive heart failure, hospitalization due to critical limb ischemia.
Frequency of indications for a second revascularization | Evaluated in 12 months from revascularization interventions
  Frequency of second revascularization events during the year.

SECONDARY OUTCOMES:
Change in the degree of stenosis of the peripheral arteries (lower limbs arteries, common carotid arteries) | Evaluated in 6 and in 12 months from revascularization interventions
  According to angiography or ultrasonography examination
Variation of intima-media thickness of common carotid arteries | Evaluated in 6 and in 12 months from revascularization interventions
  Variation of intima-media thickness of common carotid arteries measured with B-mode ultrasound of carotid arteria.
The maximal walking distance (MWD) | Evaluated in 6 and in 12 months from revascularization interventions
  Measuring the maximal walking distance (MWD) with treadmill exercise testing
Change in the ankle-brachial index (ABI) | Evaluated in 6 and in 12 months from revascularization interventions.
  Determination of the ratio systolic blood pressure within the brachial arteries and systolic blood pressure within the ankle arteries.
Change in the level of cytokine response of monocytes after double stimulation with lipopolysaccharide in in vitro cell culture | Evaluated in 6 and in 12 months from revascularization interventions
  Cytokine level measurement by ELISA (TNF-a; IL-1b; IL-6; IL-8; IL-10; CCL2) after the first and second LPS stimulation of monocytes.
Changes in the percentage of heteroplasmy of the mitochondrial genome of blood leukocytes in variants associated with atherosclerosis | Evaluated in 6 and in 12 months from revascularization interventions.
  Includes variants m.12315G>A, m.13513G>A, m.14459G>A, m.14846G>A, m.15059G>A, m.1555A>G, m.3256C>T, m.3336T>C, m.5178C>A, m.652delG measured with quantitative PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay K Shakhpazyan, PhD; Dr., Principal Investigator — "Russian research center of surgery named after academician B.V. Petrovsky"
Locations (1):
- Institute for Atherosclerosis Research, Moscow, Russia

REFERENCES:
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I, Document Reviewers, Widimsky P, Kolh P, Agewall S, Bueno H, Coca A, De Borst GJ, Delgado V, Dick F, Erol C, Ferrini M, Kakkos S, Katus HA, Knuuti J, Lindholt J, Mattle H, Pieniazek P, Piepoli MF, Scheinert D, Sievert H, Simpson I, Sulzenko J, Tamargo J, Tokgozoglu L, Torbicki A, Tsakountakis N, Tunon J, Vega de Ceniga M, Windecker S, Zamorano JL. Editor's Choice - 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2018 Mar;55(3):305-368. doi: 10.1016/j.ejvs.2017.07.018. Epub 2017 Aug 26. No abstract available. PMID 28851596
- [Background] Mahe G, Boge G, Bura-Riviere A, Chakfe N, Constans J, Goueffic Y, Lacroix P, Le Hello C, Pernod G, Perez-Martin A, Picquet J, Sprynger M; SFMV/SCVE group; SFMV/SCVE group. Disparities Between International Guidelines (AHA/ESC/ESVS/ESVM/SVS) Concerning Lower Extremity Arterial Disease: Consensus of the French Society of Vascular Medicine (SFMV) and the French Society for Vascular and Endovascular Surgery (SCVE). Ann Vasc Surg. 2021 Apr;72:1-56. doi: 10.1016/j.avsg.2020.11.011. Epub 2020 Dec 24. PMID 33359707
- [Background] Falk E. Pathogenesis of atherosclerosis. J Am Coll Cardiol. 2006 Apr 18;47(8 Suppl):C7-12. doi: 10.1016/j.jacc.2005.09.068. PMID 16631513
- [Background] Jaberi N, Soleimani A, Pashirzad M, Abdeahad H, Mohammadi F, Khoshakhlagh M, Khazaei M, Ferns GA, Avan A, Hassanian SM. Role of thrombin in the pathogenesis of atherosclerosis. J Cell Biochem. 2019 Apr;120(4):4757-4765. doi: 10.1002/jcb.27771. Epub 2018 Sep 30. PMID 30269382
- [Background] Bonati LH, Gregson J, Dobson J, McCabe DJH, Nederkoorn PJ, van der Worp HB, de Borst GJ, Richards T, Cleveland T, Muller MD, Wolff T, Engelter ST, Lyrer PA, Brown MM; International Carotid Stenting Study investigators. Restenosis and risk of stroke after stenting or endarterectomy for symptomatic carotid stenosis in the International Carotid Stenting Study (ICSS): secondary analysis of a randomised trial. Lancet Neurol. 2018 Jul;17(7):587-596. doi: 10.1016/S1474-4422(18)30195-9. Epub 2018 Jun 1. PMID 29861139
- [Background] Paraskevas KI, Giannoukas AD, Mikhailidis DP. Statins and infrainguinal vascular bypass procedures. Curr Vasc Pharmacol. 2013 Jan;11(1):51-7. PMID 23391423
- [Background] Ceyhun G, Engin MC. The Monocyte/High Density Lipoprotein Cholesterol Ratio (MHR) as an Indicator of the Need for Amputation in Patients With Peripheral Artery Disease Developing Critical Limb Ischemia. Angiology. 2021 Mar;72(3):268-273. doi: 10.1177/0003319720965808. Epub 2020 Oct 14. PMID 33108889
- [Background] Ward NC, Watts GF, Eckel RH. Response by Ward et al to Letter Regarding Article, "Statin Toxicity: Mechanistic Insights and Clinical Implications". Circ Res. 2019 Jun 7;124(12):e121-e122. doi: 10.1161/CIRCRESAHA.119.315233. Epub 2019 Jun 6. No abstract available. PMID 31170055
- [Background] Bradley JM, Organ CL, Lefer DJ. Garlic-Derived Organic Polysulfides and Myocardial Protection. J Nutr. 2016 Feb;146(2):403S-409S. doi: 10.3945/jn.114.208066. Epub 2016 Jan 13. PMID 26764335
- [Background] Orekhov AN, Tertov VV. In vitro effect of garlic powder extract on lipid content in normal and atherosclerotic human aortic cells. Lipids. 1997 Oct;32(10):1055-60. doi: 10.1007/s11745-997-0136-7. PMID 9358431
- [Background] Orekhov AN, Grunwald J. Effects of garlic on atherosclerosis. Nutrition. 1997 Jul-Aug;13(7-8):656-63. doi: 10.1016/s0899-9007(97)83010-9. PMID 9263259
- [Background] Imaizumi VM, Laurindo LF, Manzan B, Guiguer EL, Oshiiwa M, Otoboni AMMB, Araujo AC, Tofano RJ, Barbalho SM. Garlic: A systematic review of the effects on cardiovascular diseases. Crit Rev Food Sci Nutr. 2023;63(24):6797-6819. doi: 10.1080/10408398.2022.2043821. Epub 2022 Feb 23. PMID 35193446
- [Background] Mollahosseini M, Hosseini-Marnani E, Panjeshahin A, Panbehkar-Jouybari M, Gheflati A, Mozaffari-Khosravi H. A systematic review of randomized controlled trials related to the effects of garlic supplementation on platelet aggregation. Phytother Res. 2022 Nov;36(11):4041-4050. doi: 10.1002/ptr.7556. Epub 2022 Oct 12. PMID 36222178
- [Background] Panyod S, Wu WK, Chen PC, Chong KV, Yang YT, Chuang HL, Chen CC, Chen RA, Liu PY, Chung CH, Huang HS, Lin AY, Shen TD, Yang KC, Huang TF, Hsu CC, Ho CT, Kao HL, Orekhov AN, Wu MS, Sheen LY. Atherosclerosis amelioration by allicin in raw garlic through gut microbiota and trimethylamine-N-oxide modulation. NPJ Biofilms Microbiomes. 2022 Jan 27;8(1):4. doi: 10.1038/s41522-022-00266-3. PMID 35087050
- [Background] Reinhart KM, Talati R, White CM, Coleman CI. The impact of garlic on lipid parameters: a systematic review and meta-analysis. Nutr Res Rev. 2009 Jun;22(1):39-48. doi: 10.1017/S0954422409350003. PMID 19555517
- [Background] Chen ZY, Jiao R, Ma KY. Cholesterol-lowering nutraceuticals and functional foods. J Agric Food Chem. 2008 Oct 8;56(19):8761-73. doi: 10.1021/jf801566r. Epub 2008 Sep 9. PMID 18778072
- [Background] Orekhov AN, Sobenin IA, Korneev NV, Kirichenko TV, Myasoedova VA, Melnichenko AA, Balcells M, Edelman ER, Bobryshev YV. Anti-atherosclerotic therapy based on botanicals. Recent Pat Cardiovasc Drug Discov. 2013 Apr;8(1):56-66. doi: 10.2174/18722083113079990008. PMID 23176379
- [Background] Sobenin IA, Pryanishnikov VV, Kunnova LM, Rabinovich YA, Martirosyan DM, Orekhov AN. The effects of time-released garlic powder tablets on multifunctional cardiovascular risk in patients with coronary artery disease. Lipids Health Dis. 2010 Oct 19;9:119. doi: 10.1186/1476-511X-9-119. PMID 20958974
- [Background] Wlosinska M, Nilsson AC, Hlebowicz J, Hauggaard A, Kjellin M, Fakhro M, Lindstedt S. The effect of aged garlic extract on the atherosclerotic process - a randomized double-blind placebo-controlled trial. BMC Complement Med Ther. 2020 Apr 29;20(1):132. doi: 10.1186/s12906-020-02932-5. PMID 32349742
- [Background] Lindstedt S, Wlosinska M, Nilsson AC, Hlebowicz J, Fakhro M, Sheikh R. Successful improved peripheral tissue perfusion was seen in patients with atherosclerosis after 12 months of treatment with aged garlic extract. Int Wound J. 2021 Oct;18(5):681-691. doi: 10.1111/iwj.13570. Epub 2021 Feb 16. PMID 33590955
- [Background] Hamal S, Cherukuri L, Birudaraju D, Matsumoto S, Kinninger A, Chaganti BT, Flores F, Shaikh K, Roy SK, Budoff MJ. Short-term impact of aged garlic extract on endothelial function in diabetes: A randomized, double-blind, placebo-controlled trial. Exp Ther Med. 2020 Feb;19(2):1485-1489. doi: 10.3892/etm.2019.8377. Epub 2019 Dec 27. PMID 32010327
- [Background] Gao X, Xue Z, Ma Q, Guo Q, Xing L, Santhanam RK, Zhang M, Chen H. Antioxidant and antihypertensive effects of garlic protein and its hydrolysates and the related mechanism. J Food Biochem. 2020 Feb;44(2):e13126. doi: 10.1111/jfbc.13126. Epub 2019 Dec 26. PMID 31877235
- [Background] Ried K. Garlic lowers blood pressure in hypertensive subjects, improves arterial stiffness and gut microbiota: A review and meta-analysis. Exp Ther Med. 2020 Feb;19(2):1472-1478. doi: 10.3892/etm.2019.8374. Epub 2019 Dec 27. PMID 32010325
- [Background] Piragine E, Citi V, Lawson K, Calderone V, Martelli A. Potential Effects of Natural H2S-Donors in Hypertension Management. Biomolecules. 2022 Apr 14;12(4):581. doi: 10.3390/biom12040581. PMID 35454169
- [Background] Ackermann RT, Mulrow CD, Ramirez G, Gardner CD, Morbidoni L, Lawrence VA. Garlic shows promise for improving some cardiovascular risk factors. Arch Intern Med. 2001 Mar 26;161(6):813-24. doi: 10.1001/archinte.161.6.813. PMID 11268223
- [Background] Borrelli F, Capasso R, Izzo AA. Garlic (Allium sativum L.): adverse effects and drug interactions in humans. Mol Nutr Food Res. 2007 Nov;51(11):1386-97. doi: 10.1002/mnfr.200700072. PMID 17918162
- [Background] Varshney R, Budoff MJ. Garlic and Heart Disease. J Nutr. 2016 Feb;146(2):416S-421S. doi: 10.3945/jn.114.202333. Epub 2016 Jan 13. PMID 26764327